CLINICAL TRIAL: NCT00450333
Title: An Open-Label, Phase IIIb, Multi-Centre, Randomised, Parallel-Group Study to Investigate the Efficacy and Safety of Three Dosing Schedules of Subcutaneous Dynepo in Adult Patients With Anaemia Associated With Chronic Kidney Disease Who Are Pre-Dialysis or Require Peritoneal Dialysis or Haemodialysis
Brief Title: Dynepo Infrequent Dosing Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The termination of the study is not linked to a product recall or result of any safety signal. Rather it was sponsor's commercial decision to withdraw the MA
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPD490-301; 2006-002052-15 (EudraCT Number)
Record Dates: First submitted 2007-03-21; First posted 2007-03-22 (Estimated); Results first posted 2009-11-10 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Anemia; Kidney Failure
Keywords: Chronic
MeSH Terms: conditions — Anemia; Renal Insufficiency; Bronchiolitis Obliterans Syndrome | interventions — Erythropoietin; epoetin delta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Erythropoietin(EPO)-naive BIW
  Interventions: Drug: Dynepo (Epoetin delta)
- 2 (Active Comparator): EPO-naive QW
  Interventions: Drug: Dynepo
- 3 (Active Comparator): EPO QW
  Interventions: Drug: Dynepo
- 4 (Active Comparator): EPO Q2W
  Interventions: Drug: Dynepo

INTERVENTIONS:
Drug: Dynepo (Epoetin delta) — subcutaneous, BIW for 24 weeks
  Arms: 1
Drug: Dynepo — subcutaneous, QW for 24 weeks
  Arms: 2
Drug: Dynepo — subcutaneous, QW for 24 weeks
  Arms: 3
Drug: Dynepo — subcutaneous, Q2W for 24 weeks
  Arms: 4

SUMMARY:
The purpose of this study is to demonstrate non-inferiority of efficacy between twice weekly and once weekly dose schedule of Dynepo in previously erythropoietin (EPO)-naive patients, as measured by haemoglobin at week 24 and secondly to demonstrate the non-inferiority of efficacy between once weekly and once every two weeks dose schedules of Dynepo in patients previously stable on EPO, as measured by Hb over Weeks 16 to 24.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years with chronic kidney disease (Kidney Disease Outcomes Quality Initiative [KDOQI] stage III-V).
* Stable on and taking doses <= 10,000 IU/week of subcutaneous (sc) EPO or requiring initiation of EPO.
* Transferrin saturation >= 20% and ferritin >= 100 ng/mL.

Exclusion Criteria:

* Uncontrolled hypertension.
* Requiring doses of EPO > 10,000 IU/week.
* Two or more doses of prescribed EPO treatment missed ot withheld by physician order in the 14 days immediately prior tp randomisation in the study.
* Active bleeding disorder (diathesis) (for example, Gastrointestinal or Genitourinary tract bleeding).
* Treatment with immunosuppressive drugs (other than corticosteroids for a chronic condition) in the 30 days immediately prior to randomisation in the study.
* Androgen therapy in the 30 days immediately prior to randomisation in the study.
* Known Human Immunodeficiency Virus(HIV)infection.
* History of hypersensitivity to EPO therapy or to any of the excipients of Dynepo.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2006-10-30 (Actual); Primary Completion 2008-07-31 (Actual); Study Completion 2008-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (53):
- Austria (2):
  - Med.Univ-Klinik/Klin. Abt.f.Nephrologie u. Hamodialyse, Graz, Steiemark
  - Univ.-Klinik für Innere Medizin/Klin. Abt. für Nephrologie, Innsbruck
- Belgium (3):
  - Hopital UCL, Service de Nephrologie, Brussels
  - UZ Gasthuisberg, Leuve, Dept of Nephrology, Leuven
  - Hellig Hart Ziekenhuis, Campus Wilgenstraat, Roeselare
- France (10):
  - CHU - Hopital Pellegrin, Nephrologie-Hemodialyse, Bordeaux
  - CH de Boulogne-sur-mer (Hopital de Dr Duchenne), Boulogne-sur-Mer
  - Hopital Clemenceau, Nephrologie-Hemodialyse, Caen
  - CHU (Centre Hospitalier Universitaire), Grenoble
  - CHU Hotel Dieu, Service du Pr Soulillou, Nantes
  - Clinique de Landy, Service de Nephrologie - Hemodialyse, Saint-Ouen
  - Hopital Sud, Service du Pr Fournier, Salouël
  - CHU Hopital Civil, Nephrologie-Hemodialyse, Strasbourg
  - Hopital Rangueil, Service du Pr Durand, Toulouse
  - Hopital Brabois Adultes, Nephrologie, Vandœuvre-lès-Nancy
- Germany (10):
  - Nephrologische Zentrum Villingen-Schwenningen, Villingen-Schwenningen, Baden-Wurttemberg
  - KfH Nierenzentrum Bamberg, Bamberg, Bavaria
  - KfH Nierenzebtrum im Linikum Rosenheim, Rosenheim, Bavern
  - Dialyse-und Apheresezentrum Potsdam-Bebelsberg, Potsdam, Brandenburg
  - KfH Nierenzentrum Fulda, Fulda, Hesse
  - KfH Nierenzentrum am Handr-Klinikum Stralsund, Stralsund, Mecklenburg-Vorpommern
  - Gemeinschaftspraxis Prof. Mann/Prof. Heidenreich, Aachen, North Rhine-Westphalia
  - Praxis Dr. Vosskuhler, Bottrop, North Rhine-Westphalia
  - Nephrologische Gemeinschaftspraxis, Dialysezentrum Karlstrabe, Düsseldorf, North Rhine-Westphalia
  - KfK Nierenzentrum Nurnberg, Nuremberg
- Italy (10):
  - Ospedali Riuniti, Foggia, Apulia
  - Universita' degli Studi di Napoli Federico II, Napoli, Campania
  - Policlinico S. Orsola Malpighi, Bologna, Emilia-Romagna
  - Azienda Ospedaliera Universitaria Policlinico di Modena, Modena, Emillia Romagna
  - Azienda Ospedaliera S.Giovanni-Addolorata, Rome, Lazio
  - Spedali Civil Brescia, Brescia, Lombardy
  - Ospedale Nuovo Alessandro Manzoni, Lecco, Lombardy
  - Azienda Ospedaliera CTO/CRF/M.Adelaide, Turin, Piedmont
  - A.R.N.A.S Civico Palermo, Palermo, Sicily
  - Azienda Sanitaria Locale 4 Area Pratese, Prato, Tuscany
- Spain (10):
  - Hospital Puerto Real, Puerto Real, Cadiz
  - Hotel General Universitario, Castellon, Castellon
  - Head of Nephrology, Fundacion Puigvert, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Gregorio Maranon, Madrid
  - Hospital Central de Asturias, Oviedo
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Doctor Peset, Valencia
- United Kingdom (8):
  - Hope Hospital, Salford, Manchester
  - Richard Bright Renal Unit Southmead Hospital, Bristol
  - Addenbrooke's Hospital, Cambridge
  - University Hospital of Wales, Cardiff
  - Glasgow Western Infirmary, Glasgow
  - Kings College Hospital Renal Unit, London
  - Morrison Hospital, Swansea
  - New Cross Hospital, Wolverhampton

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- [Derived] Macdougall IC. Comparison of different dosing regimens (once weekly vs. twice weekly, and once weekly vs. once every two weeks) with epoetin delta in patients with chronic kidney disease: a randomized controlled trial. Trials. 2007 Nov 13;8:35. doi: 10.1186/1745-6215-8-35. PMID 17999759

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was terminated on July 31, 2008 as a result of a decision by Shire Pharmaceutical to permanently cease marketing Dynepo and withdraw the Marketing Authorisation. The decision was for commercial reasons, it was not the result of any safety signal. Not enough subjects completed the study to do any efficacy analyses.
Pre-assignment Details: Erythropoietin (EPO)-naive subjects were randomized to receive Dynepo (Epoetin delta) once weekly (QW) or twice weekly (BIW) and subjects who were already stable on EPO (doses < or equal to 10,000 IU/week) were randomized to receive Dynepo once every 2 weeks (Q2W) or once weekly.
Groups:
- Dynepo (Epoetin Delta)-Naive Once-weekly (QW): Erythropoietin(EPO)-naive subjects receiving Epoetin delta once weekly (QW)
- Dynepo-naive Twice-weekly (BIW): EPO-naive subjects receiving Epoetin delta twice weekly (BIW)
- Dynepo Once Every 2 Weeks (Q2W): EPO stable subjects receiving Epoetin delta once every 2 weeks (Q2W)
- Dynepo QW: EPO stable subjects receiving Epoetin delta once weekly (QW)
Period: Overall Study
Arm/Group | Dynepo (Epoetin Delta)-Naive Once-weekly (QW) | Dynepo-naive Twice-weekly (BIW) | Dynepo Once Every 2 Weeks (Q2W) | Dynepo QW
Started | 98 | 107 | 100 | 102
Completed | 44 | 44 | 75 | 74
Not Completed | 54 | 63 | 25 | 28
Not completed — Study terminated | 47 | 54 | 16 | 21
Not completed — Adverse Event | 1 | 7 | 2 | 2
Not completed — Protocol Violation | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 3 | 0
Not completed — Kidney transplant | 1 | 0 | 1 | 3
Not completed — Death | 3 | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dynepo (Epoetin Delta)-Naive Once-weekly (QW) | Dynepo-naive Twice-weekly (BIW) | Dynepo Once Every 2 Weeks (Q2W) | Dynepo QW | Total
Number analyzed (Participants) | 98 | 107 | 100 | 102 | 407
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 37 | 35 | 48 | 35 | 155
  >=65 years | 61 | 72 | 52 | 67 | 252
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (14.97) | 67.0 (12.45) | 64.2 (13.86) | 65.5 (16.04) | 65.7 (14.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 41 | 33 | 41 | 160
  Male | 53 | 66 | 67 | 61 | 247
Region of Enrollment [Count of Participants; unit: Participants]
  France | 6 | 8 | 8 | 3 | 25
  Spain | 3 | 2 | 13 | 14 | 32
  Belgium | 2 | 2 | 12 | 11 | 27
  Austria | 3 | 1 | 0 | 0 | 4
  Germany | 15 | 16 | 15 | 14 | 60
  United Kingdom | 10 | 15 | 11 | 12 | 48
  Italy | 5 | 5 | 28 | 35 | 73
  Australia | 19 | 22 | 7 | 6 | 54
  Hungary | 8 | 8 | 0 | 1 | 17
  Latvia | 14 | 16 | 4 | 4 | 38
  Lithuania | 10 | 9 | 0 | 0 | 19
  New Zealand | 3 | 3 | 2 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin (Hb) Concentration at 24 Weeks
Description: This study terminated early due to a decision by Shire Pharmaceuticals to permanently cease marketing Dynepo due to commercial reasons, it was not the result of any safety signal. Not enough subjects completed the study to do any efficacy analyses.
Time Frame: Baseline and 24 weeks
Population: This study terminated early due to a decision by Shire Pharmaceuticals to permanently cease marketing Dynepo due to commercial reasons, it was not the result of any safety signal. Not enough subjects completed the study to do any efficacy analyses.
Arm/Group | Dynepo (Epoetin Delta)-Naive Once-weekly (QW) | Dynepo-naive Twice-weekly (BIW) | Dynepo Once Every 2 Weeks (Q2W) | Dynepo QW
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Patients Who Achieve Hb Levels of > or Equal to 11 g/dL
Description: as for outcome 1
Time Frame: week 16 and 24
Population: as for outcome 1
Arm/Group | Dynepo (Epoetin Delta)-Naive Once-weekly (QW) | Dynepo-naive Twice-weekly (BIW) | Dynepo Once Every 2 Weeks (Q2W) | Dynepo QW
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in Hematocrits at 16 and 24 Weeks
Description: as for outcome 1
Time Frame: Baseline and Weeks 16 and 24
Population: as for outcome 1
Arm/Group | Dynepo (Epoetin Delta)-Naive Once-weekly (QW) | Dynepo-naive Twice-weekly (BIW) | Dynepo Once Every 2 Weeks (Q2W) | Dynepo QW
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Dynepo (Epoetin Delta)-Naive Once-weekly (QW) | Dynepo-naive Twice-weekly (BIW) | Dynepo Once Every 2 Weeks (Q2W) | Dynepo QW
Serious Adverse Events (participants affected / at risk) | 15/98 | 23/107 | 23/100 | 20/102
Other Adverse Events (participants affected / at risk) | 59/98 | 50/107 | 44/100 | 44/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dynepo (Epoetin Delta)-Naive Once-weekly (QW) (N=98) | Dynepo-naive Twice-weekly (BIW) (N=107) | Dynepo Once Every 2 Weeks (Q2W) (N=100) | Dynepo QW (N=102)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
DIC (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 1
Acute MI (Cardiac disorders) | 0 | 1 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 1 | 1 | 2
Peritonitis (Gastrointestinal disorders) | 3 | 0 | 1 | 2
Pneumonia (Infections and infestations) | 1 | 2 | 0 | 0
Hemoglobin decreased (Investigations) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Brain stem hemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Hypoglycemic coma (Nervous system disorders) | 0 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 2 | 2 | 2
Angina (Cardiac disorders) | 0 | 2 | 1 | 3
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Ischemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 2
Intercranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Hemorrhage (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral ischemia (Vascular disorders) | 0 | 1 | 0 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1 | 0
Duodenal ulcer hemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Intestinal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Catheter related complication (General disorders) | 0 | 0 | 1 | 0
Catheter thrombosis (General disorders) | 1 | 0 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 2 | 0
Sepsis (Infections and infestations) | 1 | 1 | 1 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 1 | 0
Arteriovenous fistula complication (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Orthopnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dynepo (Epoetin Delta)-Naive Once-weekly (QW) (N=98) | Dynepo-naive Twice-weekly (BIW) (N=107) | Dynepo Once Every 2 Weeks (Q2W) (N=100) | Dynepo QW (N=102)
Diarrhea (Gastrointestinal disorders) | 5 | 3 | 3 | 4
Nausea (Gastrointestinal disorders) | 6 | 2 | 2 | 2
Edema peripheral (General disorders) | 5 | 5 | 2 | 3
Bronchitis (Infections and infestations) | 2 | 4 | 8 | 4
Influenza (Infections and infestations) | 5 | 1 | 0 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 7 | 1 | 0 | 2
Hyperphosphatemia (Metabolism and nutrition disorders) | 5 | 5 | 3 | 1
Iron deficiency (Metabolism and nutrition disorders) | 5 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 2 | 2 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 5 | 2
Headache (Nervous system disorders) | 3 | 8 | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 5 | 3
Hypertension (Vascular disorders) | 6 | 9 | 3 | 6
Hypotension (Vascular disorders) | 1 | 2 | 5 | 3

LIMITATIONS AND CAVEATS:
This study terminated early due to a decision by Shire Pharmaceuticals to permanently cease marketing Dynepo due to commercial reasons, it was not the result of any safety signal. Not enough subjects completed the study to do any efficacy analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.